CLINICAL TRIAL: NCT01220531
Title: Safety and Efficacy of Thymus Transplantation in Complete DiGeorge Anomaly, IND#9836
Brief Title: Thymus Transplantation Safety-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00025966; 2R01AI047040-11A2 (NIH); 5K12HD043494-09 (NIH)
Record Dates: First submitted 2010-09-22; First posted 2010-10-14 (Estimated); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Complete DiGeorge Anomaly; DiGeorge Syndrome; DiGeorge Anomaly; Complete DiGeorge Syndrome
Keywords: DiGeorge Anomaly; Thymus Transplantation; DiGeorge Syndrome; Athymia; Low T cell numbers; Immunoreconstitution; Immunodeficiency; Complete DiGeorge; Typical DiGeorge; Atypical DiGeorge; Complete DiGeorge Anomaly; Cultured Thymus Tissue Implantation; Cultured Thymus Tissue; Congenital Athymia
MeSH Terms: conditions — DiGeorge Syndrome; Thymic aplasia; Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cultured Thymus Tissue (Experimental): Subjects receive thymus transplant.
  Interventions: Biological: Cultured Thymus Tissue

INTERVENTIONS:
Biological: Cultured Thymus Tissue — Potential recipients of cultured thymus tissue are screened for eligibility. The thymus tissue (from an unrelated donor), the donor, and the donor's mother are screened for safety. Cultured thymus tissue is implanted under general anesthesia in the operating room. Cultured thymus tissue is placed into the subject's quadriceps. Two to three months post-implantation, if medically stable, subjects may undergo an allograft biopsy. Subjects undergo laboratory testing for approximately one-year post-implantation. At approximately year 2 post-implantation, subjects are contacted for data collection.
  Other Names: Thymus Tissue Transplant

SUMMARY:
Complete DiGeorge anomaly (cDGA) is a disorder in which there is no thymus function. With no thymus function, bone marrow stem cells do not develop into educated T cells, which fight infection. Without successful treatment, patients with cDGA must remain in reverse isolation to prevent infection and subsequent death.

Cultured thymus tissue with and without immunosuppression (drugs given before and after implantation) has resulted in the development of good T cell function in subjects with complete DiGeorge anomaly.

This expanded access study continues cultured thymus tissue safety and efficacy research for the treatment of complete DiGeorge anomaly. Eligible participants receive cultured thymus tissue. Immune function testing is continued for one year post-implantation.

DETAILED DESCRIPTION:
Complete DiGeorge anomaly (cDGA) is a congenital disorder characterized by athymia. Without successful treatment, patients with cDGA must remain in reverse isolation to prevent infection and subsequent death. In patients with cDGA, implantation of cultured thymus tissue with and without immunosuppression has resulted in diverse T cell development and good T cell function. Protocol specified studies continue until approximately one year post-implantation. Study participation lasts two years.

Patients with Typical complete DiGeorge Anomaly usually have a) less than 50 naive T cells/mm3 or naive T cells that are less than 5% of T cells and b) a low proliferative responses to mitogens (e.g. < a 20 fold response to the mitogen phytohemagglutinin or a response of fewer than 5,000 cpm). These patients do not have diffuse rashes or lymphadenopathy. Occasional patients with typical complete DiGeorge anomaly have proliferative responses to mitogens. Patients with the typical phenotype can develop an atypical phenotype with time.

Patients with Atypical complete DiGeorge Anomaly meet the criteria for athymia (less than 50/mm3 naive T cells or less than 5% of the T cells having the naive phenotype). Patients with the atypical phenotype have developed rash, lymphadenopathy, and oligoclonal T cells. The T cells may infiltrate the liver resulting in elevated liver transaminases. The oligoclonal T cells developing in patients with DiGeorge anomaly may or may not respond to the mitogen phytohemagglutinin (PHA) in vitro.

The purpose of this expanded access study is to continue cultured thymus tissue safety and efficacy research for the treatment of athymia in patients with cDGA. Until administration of cultured thymus tissue is FDA approved as standard care for cDGA, research study participation is the only means by which a patient may have access to this potentially life-saving procedure.

This protocol includes 4 groups: one for subjects who do not require immunosuppression; and 3 immunosuppression groups for subjects with different T cell function levels to be suppressed adequately.

Group 1 :

Typical cDGA No Immunosuppression group. Subjects receive thymus transplant. Subjects do not receive any pre or post-transplantation immunosuppression.

Group 2 :

Typical and Atypical cDGA Immunosuppression group. Subjects receive thymus transplant. Subjects receive three doses of 2 mg/kg of rabbit anti-thymocyte globulin IV pre- transplantation.Medications (diphenhydramine, steroids, and acetaminophen) are given with rabbit anti-thymocyte globulin.

Group 3 :

Atypical cDGA Immunosuppression group. Subjects receive thymus transplant. Subjects receive Pre-transplant cyclosporine (Csa) as soon as complete DiGeorge anomaly is diagnosed. Csa continues with target trough levels of 180 to 220 ng/ml. When trough levels are outside of range, dosing is modified appropriately. If subject cannot tolerate Csa, the Csa may be changed to tacrolimus (FK506) with target trough level 7 to 10 ng/ml. When trough levels are outside of this target range, dosing will be modified appropriately. Pre-transplant steroids are used for atypical subjects if pre-transplant T cells >4,000/mm3. Three doses of 2 mg/kg of rabbit anti-thymocyte globulin IV are given pre-transplant. Medications (diphenhydramine, steroids, and acetaminophen) are given with rabbit anti-thymocyte globulin.

Group 4:

Atypical cDGA Additional Immunosuppression group. Subjects receive thymus transplant. Subjects receive Pre-transplant cyclosporine (Csa) and steroids are started after atypical complete DiGeorge anomaly is diagnosed. After PHA response is documented >40,000 cpm on suppression, peri-transplant Csa is maintained at target levels 250 to 300 ng/ml. (When levels outside of range, dose modified.) If subject cannot tolerate Csa then may be changed to tacrolimus (FK506) with target level 10 to 15 ng/ml. When levels are outside of range, dosing is modified. Three doses of 2 mg/kg rabbit anti-thymocyte globulin IV are given pre-transplantation. Medications (diphenhydramine, steroids, and acetaminophen) are given with rabbit anti-thymocyte globulin. Additional immunosuppression: Basiliximab, 5 mg/kg single dose IV; Mycophenolate Mofetil (MMF), 15 mg/kg/dose every 8 hours IV or enteral.

Protocol pre-specified concomitant medications

Drug: Rabbit anti-thymocyte globulin Other Names: RATGAM Three IV doses of 2 mg/kg RATGAM are given prior to implantation of cultured thymus tissue for immune suppression groups 2, 3, and 4. Each dose is given over 12 hours. RATGAM is usually given on days -5, -4, and -3 prior to implantation of cultured thymus tissue.

Drug: Cyclosporine Other Names: Csa Csa may be given every 8 or every 12 hours orally or IV before and after implantation of cultured thymus tissue for immune suppression groups 3 and 4. The Csa dose is dependent on T cell numbers and the target CSA trough levels. Csa is weaned as per protocol.

Drug: Tacrolimus Other Names: FK506 If unable to tolerate cyclosporine, then FK506 is given. FK506 may be given every 8 or every 12 hours orally or IV before and after implantation of cultured thymus tissue. FK506 dose is dependent on T cell numbers and the target FK506 trough levels. FK506 is weaned as per protocol.

Drug: Methylprednisolone or Prednisolone Other Names:Steroids Steroids IV or orally may be given before and/or after implantation of cultured thymus tissue. Steroid administration and dosage depends on T cell numbers. Steroids are weaned as per protocol.

Drug: Mycophenolate mofetil Other Names: MMF, CellCept Mycophenolate mofetil (MMF) may be given if the T cell count remains elevated 5 days after implantation of cultured thymus tissue. If MMF is given, the dose is 15 mg/kg/dose every 8 hours IV or orally. MMF may be stopped at 35 days or continued for up to six months after implantation of cultured thymus tissue.

ELIGIBILITY:
Inclusion criteria for implantation of cultured thymus tissue:

* Must have 1 of following: 22q11.2ds or 10p13 hemizygosity; hypocalcemia requiring replacement; congenital heart disease; or CHARGE syndrome or CHD7 mutation
* Complete DiGeorge: <50 CD3+ T cells/cumm or <50 CD3+ T cells/cumm that are CD62L+ CD45RA+, or <5% of CD3+ cells are CD62L+ CD45RA+
* Atypical DiGeorge subjects must have, or have had, a rash.

Group 1

•Typical cDGA whose T cells have a phytohemagglutinin (PHA) response of < 5,000 counts per minute (cpm) and < 20 fold PHA response.

Group 2

•Typical cDGA whose T cells have a PHA response of >5,000 cpm and <50,000 cpm and >20 fold PHA response.

Group 3

* Typical cDGA whose T cells have a PHA response of >50,000 cpm.
* Typical cDGA with maternal engraftment
* Atypical cDGA whose T cells have a PHA response of <40,000 cpm when on immunosuppression or <75,000 cpm to PHA when not on immunosuppression.
* Atypical cDGA with group 3 PHA response & maternal engraftment

Group 4

* Atypical cDGA with PHA responses of >75,000 cpm while on no immunosuppression or a PHA responses of >40,000 cpm while on immunosuppression.
* Atypical cDGA with maternal engraftment and group 4 PHA response

Exclusion criteria for implantation of cultured thymus tissue:

* Heart surgery conducted less than 4 weeks prior to projected implantation date.
* Heart surgery anticipated within 3 months after the proposed time of implantation
* Rejection by surgeon or anesthesiologist as surgical candidate
* Lack of sufficient muscle tissue to accept a transplant
* HIV infection
* Prior attempts at immune reconstitution, such as bone marrow transplant or previous thymus transplant
* CMV infection: For Groups 2, 3, and 4 CMV infection documented by >500 copies/ml in the blood by PCR on two consecutive assays.
* Ventilator Dependence or Positive Pressure Support: Ventilator support or positive pressure support, such as Continuous Positive Airway Pressure (CPAP) or Bi-level Positive Airway Pressure (BiPAP) support for a condition that is deemed to be severe or irreversible or which renders the subject too clinically unstable to undergo the procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Sleasman, M.D., Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology
Locations (1):
- John W. Sleasman, Durham, North Carolina, United States

REFERENCES:
- [Background] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Background] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sedlak DA, Sempowski GD, Hale LP, Rice HE, Mahaffey SM, Skinner MA. Postnatal thymus transplantation with immunosuppression as treatment for DiGeorge syndrome. Blood. 2004 Oct 15;104(8):2574-81. doi: 10.1182/blood-2003-08-2984. Epub 2004 Apr 20. PMID 15100156
- [Background] Selim MA, Markert ML, Burchette JL, Herman CM, Turner JW. The cutaneous manifestations of atypical complete DiGeorge syndrome: a histopathologic and immunohistochemical study. J Cutan Pathol. 2008 Apr;35(4):380-5. doi: 10.1111/j.1600-0560.2007.00816.x. PMID 18333898
- [Background] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Background] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Background] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Background] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sempowski GD, Rhein ME, Szabolcs P, Hale LP, Buckley RH, Coyne KE, Rice HE, Mahaffey SM, Skinner MA. Complete DiGeorge syndrome: development of rash, lymphadenopathy, and oligoclonal T cells in 5 cases. J Allergy Clin Immunol. 2004 Apr;113(4):734-41. doi: 10.1016/j.jaci.2004.01.766. PMID 15100681
- [Background] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.
- [Background] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Ciupe SM, Devlin BH, Markert ML, Kepler TB. The dynamics of T-cell receptor repertoire diversity following thymus transplantation for DiGeorge anomaly. PLoS Comput Biol. 2009 Jun;5(6):e1000396. doi: 10.1371/journal.pcbi.1000396. Epub 2009 Jun 12. PMID 19521511
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Background] Markert ML, Marques JG, Neven B, Devlin BH, McCarthy EA, Chinn IK, Albuquerque AS, Silva SL, Pignata C, de Saint Basile G, Victorino RM, Picard C, Debre M, Mahlaoui N, Fischer A, Sousa AE. First use of thymus transplantation therapy for FOXN1 deficiency (nude/SCID): a report of 2 cases. Blood. 2011 Jan 13;117(2):688-96. doi: 10.1182/blood-2010-06-292490. Epub 2010 Oct 26. PMID 20978268
- [Background] Li B, Li J, Devlin BH, Markert ML. Thymic microenvironment reconstitution after postnatal human thymus transplantation. Clin Immunol. 2011 Sep;140(3):244-59. doi: 10.1016/j.clim.2011.04.004. Epub 2011 Apr 16. PMID 21565561
- [Background] Albuquerque AS, Marques JG, Silva SL, Ligeiro D, Devlin BH, Dutrieux J, Cheynier R, Pignata C, Victorino RM, Markert ML, Sousa AE. Human FOXN1-deficiency is associated with alphabeta double-negative and FoxP3+ T-cell expansions that are distinctly modulated upon thymic transplantation. PLoS One. 2012;7(5):e37042. doi: 10.1371/journal.pone.0037042. Epub 2012 May 10. PMID 22590644
- [Background] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Background] Heimall J, Keller M, Saltzman R, Bunin N, McDonald-McGinn D, Zakai E, de Villartay JP, Moshous D, Ariue B, McCarthy EA, Devlin BH, Parikh S, Buckley RH, Markert ML. Diagnosis of 22q11.2 deletion syndrome and artemis deficiency in two children with T-B-NK+ immunodeficiency. J Clin Immunol. 2012 Oct;32(5):1141-4. doi: 10.1007/s10875-012-9741-9. Epub 2012 Aug 3. PMID 22864628
- [Background] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606
- [Background] Ciupe SM, Devlin BH, Markert ML, Kepler TB. Quantification of total T-cell receptor diversity by flow cytometry and spectratyping. BMC Immunol. 2013 Aug 6;14:35. doi: 10.1186/1471-2172-14-35. PMID 23914737
- [Background] Li B, Li J, Hsieh CS, Hale LP, Li YJ, Devlin BH, Markert ML. Characterization of cultured thymus tissue used for transplantation with emphasis on promiscuous expression of thyroid tissue-specific genes. Immunol Res. 2009;44(1-3):71-83. doi: 10.1007/s12026-008-8083-4. PMID 19066738
- [Background] Markert ML. Defects in thymic development (in Sullivan KE, Stiehm ER, eds., Stiehm's Immune Deficiencies, 2nd edition, Academic Press/Elsevier) p 357 - 379, 2020.
- [Background] Markert ML, McCarthy EA, Gupton SE, Lim AP. Cultured thymic tissue transplantation (in Sullivan KE, Stiehm ER, eds., Stiehm's Immune Deficiencies, 2nd edition, Academic Press/Elsevier) p 1229 - 1239, 2020.
- [Background] Gupton SE, McCarthy EA, Markert ML. Care of Children with DiGeorge Before and After Cultured Thymus Tissue Implantation. J Clin Immunol. 2021 Jul;41(5):896-905. doi: 10.1007/s10875-021-01044-0. Epub 2021 May 18. PMID 34003433
- [Background] Markert ML, Gupton SE, McCarthy EA. Experience with cultured thymus tissue in 105 children. J Allergy Clin Immunol. 2022 Feb;149(2):747-757. doi: 10.1016/j.jaci.2021.06.028. Epub 2021 Aug 4. PMID 34362576

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cultured Thymus Tissue
Started | 29
Completed | 21
Not Completed | 8
Not completed — Death | 7
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cultured Thymus Tissue
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: Days] | 449.7 (226.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 21
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at End of 1 Year
Time Frame: 1 year
Population: Efficacy Analysis Set (EAS): EAS set includes all subjects with athymia associated with complete DiGeorge anomaly or FoxN1 deficiency, who had no prior hematopoietic cell transplant (HCT) and were treated with cultured postnatal thymus tissue in study 25966
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cultured Thymus Tissue
Number analyzed (Participants) | 29
percentage of participants | 79.3 [60 to 92]

2. Primary Outcome: Survival Rate at End of 2 Year
Time Frame: 2 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cultured Thymus Tissue
Number analyzed (Participants) | 29
percentage of participants | 75 [55 to 89]

ADVERSE EVENTS:
Time Frame: 2 Years
Description: within 2 Years of Transplantation
Arm/Group | Cultured Thymus Tissue
All-Cause Mortality (participants affected / at risk) | 7/29
Serious Adverse Events (participants affected / at risk) | 24/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue (N=29)
Device related infection (Infections and infestations) | 14 (33)
Lower respiratory tract infection bacterial (Infections and infestations) | 3 (4)
Pneumonia (Infections and infestations) | 3 (3)
Klebsiella bacteraemia (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pyrexia (General disorders) | 7 (8)
Pancreatitis (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 2 (2)
Graft versus host disease (Immune system disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue (N=29)
Viral upper respiratory tract infection (Infections and infestations) | 7 (7)
Device related infection (Infections and infestations) | 6 (8)
Oropharyngeal candidiasis (Infections and infestations) | 6 (7)
Lower respiratory tract infection bacterial (Infections and infestations) | 4 (9)
Pneumonia (Infections and infestations) | 4 (4)
Enterobacter pneumonia (Infections and infestations) | 3 (3)
Fungal skin infection (Infections and infestations) | 3 (3)
Gastroenteritis norovirus (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Urinary tract infection bacterial (Infections and infestations) | 3 (7)
Bacterial tracheitis (Infections and infestations) | 2 (4)
Klebsiella bacteraemia (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 2 (2)
Sinusitis bacterial (Infections and infestations) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 2 (3)
Stoma site infection (Infections and infestations) | 2 (2)
Viraemia (Infections and infestations) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 5 (5)
Splenomegaly (Blood and lymphatic system disorders) | 2 (2)
Cytokine release syndrome (Immune system disorders) | 5 (5)
Hypothyroidism (Endocrine disorders) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Cardiomegaly (Cardiac disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (6)
Thrombosis (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (9)
Haematochezia (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 13 (19)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Pyrexia (General disorders) | 12 (17)
Granuloma (General disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Alanine aminotransferase increased (Investigations) | 5 (7)
Blood creatinine increased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT01220531/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT01220531/SAP_001.pdf